CLINICAL TRIAL: NCT03416387
Title: Single Arm Trial of Applicability of 3D Printing and 3D Digital Image Reconstruction in the Planning of Complex Liver Surgery.
Brief Title: Applicability of 3D Printing and 3D Digital Image Reconstruction in the Planning of Complex Liver Surgery (LIV3DPRINT).
Acronym: LIV3DPRINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Ricardo Robles Campos, Profesor, Hospital Universitario Virgen de la Arrixaca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LIV3DPRINT
Record Dates: First submitted 2017-12-19; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Liver Diseases; Surgery
Keywords: complex liver surgery; 3D printing
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OTHER: 3D PRINTING AND 3D DIGITAL IMAGE RECONSTRUCTION (Other)
  Interventions: Device: 3D PRINTING

INTERVENTIONS:
Device: 3D PRINTING — A 3D digital image reconstruction and a 3D printing model were performed in all patients with complex liver tumors.

SUMMARY:
Three-dimensional (3D) printing has gained popularity in medicine over the last decade. Once 3D printers have become more affordable, the true strength of this technique has been recognized because of its ability to obtain anatomical models based on the unique characteristics of each patient. Liver resections are challenging operations because of the complex nature of the liver and venous anatomy within the liver, so 3D imaging is a promising new tool for surgical planning.

ELIGIBILITY:
Inclusion Criteria:

* Complex liver tumors (bilobar disease, infiltration of suprahepatic veins or requiring two-time resection or intrahepatic vascular reconstruction).
* Preoperatively was performed, a CT scan and / or MRI of all patients were performed to document the tumor distribution, estimate remaining liver volume, and identify tumor-vessel relationships in order to know the intraoperative vascular anatomy.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-23 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Surgical planing | 2 weeks
  Number of Participants susceptible of complex liver surgery as assessed by 3D printing and 3D digital image reconstruction, change from the baseline to the surgical strategy

SECONDARY OUTCOMES:
Teaching for students and residents | 1 day
  Number of students where 3D models of digital printing and images reconstructed in 3D by using a questionnaire improve understanding about the location of lesions, liver anatomy and planning of surgery
Understanding of surgery by the patient | 1day
  Number of patient who understand better liver disease and surgery strategy

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic and University Virgen de la Arrixaca Hospital, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Good practice principles include: (i) the use of a controlled access approach, using a transparent and robust system to review requests and provide secure data access; (ii) seeking consent for sharing IPD from trial participants in all future clinical trials with adequate assurance that patient privacy and confidentiality can be maintained; and (iii) establishing an approach to resource the sharing of IPD which would include support from trial funders, sponsor organisations and users of IPD.